CLINICAL TRIAL: NCT05602467
Title: Efficacy of a 24-week Long Term Transcranial Pulse Stimulation (TPS) on Cognition and Brain Structure in Older Adults With Mild Neurocognitive Disorder (NCD)
Brief Title: Long Term Transcranial Pulse Stimulation (TPS) on Older Adults With Mild Neurocognitive Disorder (NCD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Storz Medical AG (Industry)
Responsible Party: Principal Investigator, Dr. Cheng Pak Wing, Calvin, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW22-642
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Mild Neurocognitive Disorder
Keywords: TPS; Transcranial Pulse Stimulation; Mild Neurocognitive Disorder; Open-Label; long term intervention
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Transcranial Magnetic Stimulation; Therapeutics

STUDY DESIGN:
Intervention Model Description: The active group would receive 2 stimulation programs, each set last 12-week. Participants would receive 3 sessions/week in the first 2 weeks and then 1 session/week in the subsequent 10 weeks. A total of 32 sessions (16 sessions per set) of TPS will be delivered, each lasting 30 minutes.
  The control group will be recruited with the same recruitment criteria. They would receive treatment-as-usual (TAU) in the outpatient clinic without TPS intervention given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): A total of 32 sessions (2 sets of 16 sessions) of TPS will be delivered, each lasting 30 minutes. Each set includes 3 sessions per week in the first 2 weeks and then 1 session per week in the subsequent 10 weeks.
  Interventions: Device: Transcranial Pulse Stimulation (TPS)
- Control Group (Placebo Comparator): The control group will be recruited with the same recruitment criteria. They would receive treatment-as-usual (TAU) in the outpatient clinic without TPS intervention given.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Device: Transcranial Pulse Stimulation (TPS) — A global brain stimulation approach, which homogenously distributes the total energy of 6000 TPS pulses per session over all accessible brain areas.
  Prefrontal, Temporal and Occipital brain areas were stimulated by ultrashort (3μs) ultrasound pulses with typical energy levels of 0.2-0.25 mJ/mm2 and pulse frequencies of 4-5 Hz (pulses per second).
  Arms: Treatment Group
Other: Treatment as usual (TAU) — Treatment-as-usual (TAU) in the Hong Kong outpatient clinic without TPS intervention was given. They would receive the standard care for mild NCD including counselling, lifestyle modification, cognitive training and antidementia medications occasionally depending on the case doctor's judgement.
  Arms: Control Group

SUMMARY:
Background:

Dementia, now known as major neurocognitive disorder (NCD), is a great health burden in Hong Kong and worldwide. In principle, to achieve its optimal benefits, intervention for dementia should begin at the earliest preclinical stage, which is defined as mild cognitive impairment (MCI). However, no evidence has been found to support a pharmacological approach to the prevention or postponement of cognitive decline during the stage of mild NCD. Non-invasive brain stimulation (NIBS) is increasingly recognized as a potential alternative to tackle this problem.

The typical examples of NIBS are transcranial direct current stimulation (DCS) and transcranial magnetic stimulation (MS). Besides these, there is a new NIBS named transcranial pulse stimulation (TPS), which recently obtained CE marking in 2018 for the treatment of the central nervous system (CNS) in patients with mild to moderate Alzheimer's disease (AD). TPS is using repetitive single ultrashort pulses in the ultrasound frequency range to stimulate the brain. With a neuro-navigation device, TPS can achieve this in a highly focal and precisely targeted manner. TPS differs from DCS and TMS using direct or induced electric current. Instead, TPS provides good spatial precision and resolution to noninvasively modulate subcortical areas, despite the problem of skull attenuation. Using lower ultrasound frequencies TPS can successfully improve skull penetration in humans. TPS has shown its neuroprotective effects through inducing long term neuroplastic changes, supported by neuropsychological tests and neuroimaging investigations both in animal and human studies.

Mild NCD is a golden period for intervention to avoid further progression to dementia. Although TPS has great potential as a new treatment option due to its neuroprotective effects, there is no TPS study done on mild CD subjects according to our knowledge. To determine the effectiveness of TPS in mild NCD, an open-label pilot study was conducted by our team from Dec 2020 to Dec 2021. The preliminary result was presented in the 2021 Brain Stimulation Conference and published in abstract format. We recruited 16 older adults who had mild CD. They received 6 sessions of TPS over 2 weeks.

Assessments were done at the 3 time points. No subjects dropped out during the study. Statistically significant improvement was found in the primary outcome, HK-MoCA, from 18.06 to 20.25. The improvement was maintained till 12 weeks after the TPS intervention. No adverse effect was observed. The result suggested that TPS is likely to have an immediate effect on global cognition in mild CD, and the improvements were sustainable. However, a 2-week treatment duration may not be long enough to induce a significant change in neurodegenerative disease in long term. Up to date, there is no long-term NIBS treatment done on NCD. Therefore, we plan to conduct a pilot case-controlled trial to evaluate the efficacy of long-term TPS on cognition and brain structure in patients with mild ND based on the results of our pilot study.

Objective:

This study is to determine the efficacy of a 24-week program (32 sessions) of TPS in older adults with mild NCD. We hypothesized that TPS group is significantly more effective than control group in maintain or improve the global cognitive function measured by Hong Kong Chinese version of Montreal Cognitive Assessment (HK-MoCA) in patients with mild NCD.

Design:

This case-controlled trial will assess the efficacy of a 24-week TPS program on cognition and brain structure in subjects with mild NCD. All eligible participants will receive an intervention trial of TPS. They would receive 2 sets of stimulation programs, each set lasting 12-weeks. Participants would receive 3 sessions/week in the first 2 weeks and then 1 session/week in the subsequent 10 weeks. A total of 32 sessions (2 sets of 16 sessions) ofTPS will be delivered, with each session lasting 30 minutes.

Data Analysis:

The primary and secondary outcomes will be assessed at baseline, immediately after the 1st set of stimulation program (12th week), 2nd set of stimulation program (24th week), and 12 weeks after the intervention (36th week). The primary outcome will be the change of the Hong Kong Chinese version of the Montreal Cognitive Assessment (HK-MoCA). The secondary outcome includes specific cognitive domains, daily functioning, mood, and apathy. The intention-to-treat analysis would be carried out. Pre and post-intervention brain MRI scans will be used during the intervention to evaluate the changes in brain structure. A checklist of potential adverse effects associated with TPS administration will be generated from the available literature. Blood pressure and heart rate will be recorded at the beginning and at the end of the TPS intervention course.

DETAILED DESCRIPTION:
Background:

Dementia, now known as major neurocognitive disorder (NCD), is a great health burden in Hong Kong and worldwide. Interventions that aim to ameliorate cognitive decline or prevent dementia offer a compelling alternative paradigm for reducing the impact of the disease. In principle, to achieve its optimal benefits, intervention for dementia should begin at the earliest preclinical stage, which is defined as mild cognitive impairment (MCI) or mild NCD defined by the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

However, no evidence has been found to support a pharmacological approach to the prevention or postponement of cognitive decline during the stage of mild NCD or MCI (1, 2). Non-invasive brain stimulation (NIBS) is increasingly recognized as a potential alternative to tackle this problem.

The introduction of TPS:

The typical examples of NIBS are transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS). Besides these, there is a new NIBS named transcranial pulse stimulation (TPS), which recently obtained CE marking in 2018 for the treatment of the central nervous system (CNS) in patients with mild to moderate Alzheimer's disease (AD).

TPS is using repetitive single ultrashort pulses in the ultrasound frequency range to stimulate the brain. With a neuro-navigation device, TPS can achieve this in a highly focal and precisely targeted manner (3). TPS differs from tDCS and TMS using direct or induced electric current. Using electric current to stimulate the brain may be limited by the problem of conductivity (4) and failure to reach deep brain regions (5). Instead, TPS provides good spatial precision and resolution to noninvasively modulate subcortical areas, despite the problem of skull attenuation (6). Using lower ultrasound frequencies TPS can successfully improve skull penetration in humans (3).

Biological mechanism of TPS:

The basic mechanism of TPS is mechanotransduction. It is a biological pathway through which the cells convert the mechanical TPS stimulus into biochemical responses, thus influencing some fundamental cell functions such as migration, proliferation, differentiation, and apoptosis (7, 8). The ultrashort ultrasound pulse could enhance cell proliferation and differentiation in cultured neural stem cells, which plays an important role in the repair of brain function in CNS diseases (9). The TPS probably affects neurons and induces neuroplastic effects through several pathways including increasing cell permeability (9), stimulation of mechanosensitive ion channels (7), the release of nitric oxide resulting in vasodilation, increased metabolic activity and angiogenesis (10), stimulation of vascular growth factors (VEGF) (11) and stimulation of brain-derived neurotrophic factor (BDNF) (12). Another animal study showed that ultrasound stimulation immediately after ischemic brain injury is neuroprotective through the increase of cerebral blood flow and activation of the synthesis of nitric oxide (13).

Previous clinical experience of TPS and its safety issue:

TPS demonstrated neuromodulation effects in the human brain. There are a few advantages of TPS techniques. First, the ultrashort TPS pulses avoid brain heating and secondary stimulation maxima. Second, TPS can modulate the amplitude of somatosensory evoked potentials (SEPs) at both the cortical regions (3) and even the deep structure such as the thalamus (6). Third, TPS may alter human brain morphology (14).

For clinical use, long-term TPS was shown to bring significant improvement in patients with unresponsive wakefulness syndrome. (15). In another clinical study, TPS was applied to elderly with AD. Significant improvement in cognition was demonstrated (immediately as well as 1 and 3 months after stimulation. fMRI also showed significantly increased connectivity within the memory network (3). During the subsequent follow-up in the same study, TPS has been shown reduced cortical atrophy within the default mode network, which is associated with neuropsychological improvement (14). Another TPS study done on the human brain found that the active TPS increased the functional and structural coupling within the stimulated area and adjacent areas up to one week after the last stimulation compared with the sham TPS control. It suggested that TPS could induce neuroplastic changes with long-term effects in humans (16). In summary, TPS has shown its neuroprotective effects by inducing long-term neuroplastic changes, supported by neuropsychological tests and neuroimaging investigations both in animal and human studies.

Concerning the safety issue, in vivo animal TPS study did not cause any tissue damage despite using 6-7-fold higher energy levels compared with those in human studies. Furthermore, the intervention did not cause any serious adverse effects such as intracranial bleeding, oedema or other intracranial pathology in human, as confirmed with MRI in a previous AD study. No serious adverse effects except headache (4%), pain or pressure (1%) and mood deterioration (3%) was reported (3). The CE marked TPS system has proven to be safe in >1500 treatments.

Knowledge gap and results from our pilot study:

Mild NCD is a golden period for intervention to avoid further progression to dementia. Although TPS has great potential as a new treatment option due to its neuroprotective effects, there is no TPS study done on mild NCD subjects according to our knowledge. To determine the effectiveness of TPS in mild NCD, an open-label pilot study was conducted by our team from Dec 2020 to Dec 2021. (Appendix 1) The preliminary result was presented at 2021 Brain Stimulation Conference and published in abstract format (17). We recruited 16 older adults who had mild NCD. They received 6 sessions of TPS over 2 weeks. Assessments were done at the 3 time points. No subjects dropped out during the study. Statistically significant improvement was found in the primary outcome, HK-MoCA, from 18.06 to 20.25. The improvement was maintained till 12 weeks after the TPS intervention. No adverse effect was observed. The result suggested that TPS is likely to have an immediate effect on global cognition in mild NCD, and the improvements were sustainable. However, a 2-week treatment duration may not be long enough to induce a significant change in neurodegenerative disease in long term. Previous research showed that long-term deep brain stimulation may reverse hippocampal atrophy and influence the natural course of brain atrophy in Alzheimer's disease (AD) (18). Up to date, there is no long-term NIBS treatment done on NCD. Therefore, we plan to conduct a pilot case-controlled trial to evaluate the efficacy of long-term TPS on cognition and brain structure in patients with mild NCD based on the results of our pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years of age or above
2. Chinese ethnicity
3. Fulfil the criteria of mild neurocognitive disorder (NCD), defined by the DSM-5
4. Stable dosage/frequency of anti-dementia therapy or other treatments for mild NCD in recent 8 weeks
5. Valid informed written consent

Exclusion Criteria:

1. HK-MoCA score below the second percentile according to the subject's age and education level (to exclude subjects with existing major NCD/dementia)
2. Alcohol or substance dependence
3. Concomitant unstable major medical conditions or major neurological conditions such as brain tumour, recent stroke
4. Haemophilia or other blood clotting disorders or thrombosis
5. Significant communicative impairments
6. Participants with any metal implant in brain or treated area of the head

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in Global Cognition | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Global cognitive function measured by the Hong Kong Chinese version of the Montreal Cognitive Assessment (HK-MoCA) ranges from 0 to 30, with higher scores indicating better cognition.

SECONDARY OUTCOMES:
Change in Memory | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Measured by Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) - Chinese version
Change in Executive Function | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Measured by Stroop test.
Change in Attention/Working Memory | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Measured by Trail Making Test Parts A and B
Change in Brain Structure | Baseline, 12-week Follow-up
  Structural MRI will be performed using a 3T scanner at HKU. Pre and post intervention brain MRI scan will be used during intervention and evaluate the changes in brain structure. The participants' brain images will be loaded into the TPS machine before the session start. Those participants with abnormal brain scan result such as brain tumour and recent stroke will be excluded. Images processing and analysis will be performed using software packages including FSL and SPM8 to assess the voxel-based morphometry (VBM) in hippocampus and other relevant regions.
Change in Daily Functioning | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Measured by Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living Scale.
Change in Mood | Baseline, at 12 weeks, at 24 weeks, 12-week Follow-up
  Measured by the Depression Rating Scale (HAMD-17)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin PW Cheng, MBBS (HKU), Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Jockey Club Building for Interdisciplinary Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Since the study involves sensitive and private medical history from recruited or self-enrolled subjects, individual data will not be available to other researchers.

REFERENCES:
- [Background] Cooper C, Li R, Lyketsos C, Livingston G. Treatment for mild cognitive impairment: systematic review. Br J Psychiatry. 2013 Sep;203(3):255-64. doi: 10.1192/bjp.bp.113.127811. PMID 24085737
- [Background] Kasper S, Bancher C, Eckert A, Forstl H, Frolich L, Hort J, Korczyn AD, Kressig RW, Levin O, Palomo MSM. Management of mild cognitive impairment (MCI): The need for national and international guidelines. World J Biol Psychiatry. 2020 Oct;21(8):579-594. doi: 10.1080/15622975.2019.1696473. Epub 2020 Feb 5. PMID 32019392
- [Background] Beisteiner R, Matt E, Fan C, Baldysiak H, Schonfeld M, Philippi Novak T, Amini A, Aslan T, Reinecke R, Lehrner J, Weber A, Reime U, Goldenstedt C, Marlinghaus E, Hallett M, Lohse-Busch H. Transcranial Pulse Stimulation with Ultrasound in Alzheimer's Disease-A New Navigated Focal Brain Therapy. Adv Sci (Weinh). 2019 Dec 23;7(3):1902583. doi: 10.1002/advs.201902583. eCollection 2020 Feb. PMID 32042569
- [Background] Minjoli S, Saturnino GB, Blicher JU, Stagg CJ, Siebner HR, Antunes A, Thielscher A. The impact of large structural brain changes in chronic stroke patients on the electric field caused by transcranial brain stimulation. Neuroimage Clin. 2017 Apr 18;15:106-117. doi: 10.1016/j.nicl.2017.04.014. eCollection 2017. PMID 28516033
- [Background] Spagnolo PA, Wang H, Srivanitchapoom P, Schwandt M, Heilig M, Hallett M. Lack of Target Engagement Following Low-Frequency Deep Transcranial Magnetic Stimulation of the Anterior Insula. Neuromodulation. 2019 Dec;22(8):877-883. doi: 10.1111/ner.12875. Epub 2018 Oct 29. PMID 30370983
- [Background] Legon W, Ai L, Bansal P, Mueller JK. Neuromodulation with single-element transcranial focused ultrasound in human thalamus. Hum Brain Mapp. 2018 May;39(5):1995-2006. doi: 10.1002/hbm.23981. Epub 2018 Jan 29. PMID 29380485
- [Background] d'Agostino MC, Craig K, Tibalt E, Respizzi S. Shock wave as biological therapeutic tool: From mechanical stimulation to recovery and healing, through mechanotransduction. Int J Surg. 2015 Dec;24(Pt B):147-53. doi: 10.1016/j.ijsu.2015.11.030. Epub 2015 Nov 28. PMID 26612525
- [Background] Ingber DE. Cellular mechanotransduction: putting all the pieces together again. FASEB J. 2006 May;20(7):811-27. doi: 10.1096/fj.05-5424rev. PMID 16675838
- [Background] Zhang J, Kang N, Yu X, Ma Y, Pang X. Radial Extracorporeal Shock Wave Therapy Enhances the Proliferation and Differentiation of Neural Stem Cells by Notch, PI3K/AKT, and Wnt/beta-catenin Signaling. Sci Rep. 2017 Nov 10;7(1):15321. doi: 10.1038/s41598-017-15662-5. PMID 29127399
- [Background] Mariotto S, Cavalieri E, Amelio E, Ciampa AR, de Prati AC, Marlinghaus E, Russo S, Suzuki H. Extracorporeal shock waves: from lithotripsy to anti-inflammatory action by NO production. Nitric Oxide. 2005 Mar;12(2):89-96. doi: 10.1016/j.niox.2004.12.005. PMID 15740982
- [Background] Hatanaka K, Ito K, Shindo T, Kagaya Y, Ogata T, Eguchi K, Kurosawa R, Shimokawa H. Molecular mechanisms of the angiogenic effects of low-energy shock wave therapy: roles of mechanotransduction. Am J Physiol Cell Physiol. 2016 Sep 1;311(3):C378-85. doi: 10.1152/ajpcell.00152.2016. Epub 2016 Jul 13. PMID 27413171
- [Background] Wang B, Ning H, Reed-Maldonado AB, Zhou J, Ruan Y, Zhou T, Wang HS, Oh BS, Banie L, Lin G, Lue TF. Low-Intensity Extracorporeal Shock Wave Therapy Enhances Brain-Derived Neurotrophic Factor Expression through PERK/ATF4 Signaling Pathway. Int J Mol Sci. 2017 Feb 16;18(2):433. doi: 10.3390/ijms18020433. PMID 28212323
- [Background] Guo T, Li H, Lv Y, Lu H, Niu J, Sun J, Yang GY, Ren C, Tong S. Pulsed Transcranial Ultrasound Stimulation Immediately After The Ischemic Brain Injury is Neuroprotective. IEEE Trans Biomed Eng. 2015 Oct;62(10):2352-7. doi: 10.1109/TBME.2015.2427339. Epub 2015 Apr 28. PMID 25935023
- [Background] Lohse-Busch H, Reime U, Falland R. Symptomatic treatment of unresponsive wakefulness syndrome with transcranially focused extracorporeal shock waves. NeuroRehabilitation. 2014 Jan 1;35(2):235-44. doi: 10.3233/NRE-141115. PMID 24990026
- [Background] Matt E, Kaindl L, Tenk S, Egger A, Kolarova T, Karahasanovic N, Amini A, Arslan A, Saricicek K, Weber A, Beisteiner R. First evidence of long-term effects of transcranial pulse stimulation (TPS) on the human brain. J Transl Med. 2022 Jan 15;20(1):26. doi: 10.1186/s12967-021-03222-5. PMID 35033118
- [Background] Sankar T, Chakravarty MM, Bescos A, Lara M, Obuchi T, Laxton AW, McAndrews MP, Tang-Wai DF, Workman CI, Smith GS, Lozano AM. Deep Brain Stimulation Influences Brain Structure in Alzheimer's Disease. Brain Stimul. 2015 May-Jun;8(3):645-54. doi: 10.1016/j.brs.2014.11.020. Epub 2014 Dec 3. PMID 25814404
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Lam LC, Tam CW, Lui VW, Chan WC, Chan SS, Chiu HF, Leung T, Tham MK, Ho KS, Chan WM. Screening of mild cognitive impairment in Chinese older adults--a multistage validation of the Chinese abbreviated mild cognitive impairment test. Neuroepidemiology. 2008;30(1):6-12. doi: 10.1159/000113300. Epub 2008 Jan 17. PMID 18204291
- [Background] Farrer LA, Cupples LA, Haines JL, Hyman B, Kukull WA, Mayeux R, Myers RH, Pericak-Vance MA, Risch N, van Duijn CM. Effects of age, sex, and ethnicity on the association between apolipoprotein E genotype and Alzheimer disease. A meta-analysis. APOE and Alzheimer Disease Meta Analysis Consortium. JAMA. 1997 Oct 22-29;278(16):1349-56. PMID 9343467
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Zheng YP, Zhao JP, Phillips M, Liu JB, Cai MF, Sun SQ, Huang MF. Validity and reliability of the Chinese Hamilton Depression Rating Scale. Br J Psychiatry. 1988 May;152:660-4. doi: 10.1192/bjp.152.5.660. PMID 3167442
- See also: Cheng PWC, Fong KHT. Efficacy and safety of transcranial pulse stimulation (TPS) in older adults with mild neurocognitive disorder-an open-label trial. Brain Stimulation: Basic, Translational, and Clinical Research in Neuromodulation. 2021;14(6):1636. — https://doi.org/10.1016/j.brs.2021.10.155